CLINICAL TRIAL: NCT01439217
Title: Endothelial Function, Arterial Stiffness and Components of Metabolic Syndrome in Acute Lymphoblastic Leukemia (ALL) Survivors
Brief Title: Endothelial Function, Arterial Stiffness and Components
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J1064; NA_00040838 (Other: JHMIRB)
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; Survivor; Sibling control
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Specific Aim: Compare the endothelial function, arterial stiffness and components of metabolic syndrome of childhood Acute Lymphoblastic Leukemia (ALL) survivors to healthy sibling controls. Plan: A cross sectional study comparing ALL survivors to sibling controls including measures of endothelial function and arterial stiffness obtained form a peripheral artery tonometry device, height, weight, waist circumference, fasting lipid, glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

Survivor:

Inclusion

1. Ages 8-28 (8 is chosen as lower age limit because developmental understanding will allow survivor to follow instructions for procedures, 28 is chosen as upper limit to include age ranges seen for treatment in the pediatric program)
2. Off therapy for at least 6 months and not more than 10 years (6 months

Inclusion

1. Biological sibling
2. Ages 8-28 (when more than one sibling is available the one closest in age will be chosen.))

Exclusion Criteria:

1. Uncontrolled medical conditions that could interfere with participation or interpretation of results
2. History of relapsed ALL or history of bone marrow transplantation

Ages: 8 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This descriptive, healthy sibling control study will utilize a convenience sample of 20 childhood ALL survivors, recruited from the Survivorship Program at Johns Hopkins (SPJH). The study will be introduced to survivors/parent/guardians during routine clinic visits. If they are interested in participation the consent form for both the survivor and sibling will be reviewed and taken home to discuss with the sibling and other family members. Follow-up phone call and questions will be encouraged. If all parties agree to participate an appointment will be set up to enroll the survivor/sibling and face to face informed consent will be obtained.
  A second method for recruitment will include mailings (see attached) to ALL survivors seen/treated at Johns Hopkins. Letters will include phone and email contacts to acquire further information and a post card to decline further contact.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
measure of endothelial | at enrollment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland